CLINICAL TRIAL: NCT05594537
Title: The Best Way to Improve the Near Visual Acuity After Implantation of Tecnis Symfony® ZXR00 Intraocular Lens
Brief Title: The Best Way to Improve the Near Visual Acuity After ZXR00 IOL Implantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: ZXR00-zyy
Record Dates: First submitted 2022-10-20; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cataract; Near Vision
MeSH Terms: conditions — Cataract; Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ZXR00+ZXR00 emmetropia group: The bilateral implantation of ZXR00 IOLs，and emmetropia was considered as the target refraction for both eyes.
- ZXR00+ZXR00 micromonovision group: The bilateral implantation of ZXR00 IOLs，and the ZXR00 IOLs power calculations were performed using a micro-monovision approach aiming for minimal residual myopia (≈ -0.50 D) in the nondominant eye and emmetropia in the dominant eye.
- ZXR00ZMB00 group: The blended implantation of bifocal IOLs (ZMB00) and ZXR IOLs.

SUMMARY:
The Best Way to Improve the Near Visual Acuity After ZXR00 IOL Implantation

DETAILED DESCRIPTION:
ZXR00 intraocular lens is a new type of IOL that can achieve good continuous visual acuity. Its characteristic is to improve the distance and intermedia visual acuity and maintain good visual quality while sacrificing the near visual acuity. Previous studies report that there are mainly two ways to improve the near visual acuity of ZXR00：1.Bilateral implantation of ZXR00 with micromonovision. 2. Combined Implantation of ZXR00 and multifocal IOLs.This study aim to explore which is the best way to improve the near visual acuity after ZXR00 IOL implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-80 years
* Cataract surgery is planned
* The operation was successful without any complications
* Implanted with ZXR00 IOLS or ZMB00 IOLs

Exclusion Criteria:

* The history of retinopathy or retinal surgery
* Irregular corneal astigmatism
* Regular corneal astigmatism of 1.00 diopter (D) or more
* Iris abnormalities
* Macular degeneration
* Neuro-ophthalmic disease
* The history of ocular inflammation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From December 2019 to present, cataract patients underwent phacoemulsification combined with ZXR00 IOLs or ZMB00 IOLs implantation by an experienced ophthalmologist (Dr. Zhao Yune) in Wenzhou Medical University Affiliated Eye Hospital(hangzhou branch).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Visual Acuities | 2022.12.31
  Uncorrected monocular and binocular visual acuities (logarithm of the minimum angle of resolution) at distance (5m), intermediate(66 cm), and near (40 cm).
Corrected Visual Acuities | 2022.12.31
  Corrected monocular and binocular visual acuities (logarithm of the minimum angle of resolution) at distance (5m), intermediate(66 cm), and near (40 cm).
Defocus Curve | 2022.12.31
  Corrected monocular and binocular defocus curves were measured from +2.5 D to -4.0 D (in 0.5 D steps).
Patient satisfaction | 2022.12.31
  Patient satisfaction was rated on a scale of 1 to 5: 1 = very dissatisfied; 2 = dissatisfied; 3 = neutral; 4 = satisfied; and 5 = very satisfied.
Subjective quality of vision | 2022.12.31
  Subjective quality of vision was evaluated using the 14-item Visual Function Questionnaire (VFQ-14).Each item was scaled according to the degree of difficulty of different activities: 4 points (no difficulty), 3 points (a little difficulty), 2 points (a moderate amount of difficulty), 1 point (a great deal of difficulty), and 0 point (unable to do the activity).overall score is range 0-56.The higher the score, the worse subjective quality of vision.
Adverse visual symptoms | 2022.12.31
  Adverse visual symptoms including blurred vision, glare, starbursts, haloes, hazy vision, distortion, focusing diffculties, multiple images, and depth perception diffculty, was evaluated using the Quality of Vision test. This test includes 30 items, with a score between 0 and 3 (overall score range 0-90).The higher the score, the more postoperative adverse visual symptoms.
Stereopsis | 2022.12.31
  Stereopsis was evaluated using OCULUS Binoptometer.

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Ophthalmology and Optometry Hospital